CLINICAL TRIAL: NCT00677118
Title: A Multicenter Prospective Randomized Trial Comparing Concurrent Chemoradiotherapy Plus Adjuvant Chemotherapy With Concurrent Chemoradiotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Adjuvant Chemotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other); Zhejiang Cancer Hospital (Other); Huazhong University of Science and Technology (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Peking University Cancer Hospital & Institute (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Jun Ma, Sun Yat-sen University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YP2008004
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2010-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Concurrent chemoradiotherapy; Adjuvant chemotherapy; Clinical trial
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — CF regimen; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent and adjuvant (Experimental): Concurrent chemoradiotherapy plus adjuvant chemotherapy
  Interventions: Drug: Cisplatin,fluorouracil
- Concurrent (Active Comparator): Concurrent chemoradiotherapy
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin,fluorouracil — Patients receive radical radiotherapy and cisplatin (40mg/m2 on day 1) weekly during radiotherapy, then receive cisplatin (80mg/m2 on day 1) and fluorouracil (800mg/m2 on Day 1 to 5) every four weeks for three cycles after completion of radiotherapy.
  Other Names: Cisplatin and fluorouracil
  Arms: Concurrent and adjuvant
Drug: Cisplatin — Patients receive radical radiotherapy and cisplatin (40mg/m2 on day 1) weekly during radiotherapy.
  Arms: Concurrent

SUMMARY:
The purpose of this study is to compare concurrent chemoradiotherapy plus adjuvant chemotherapy with concurrent chemoradiotherapy in patients with locoregionally advanced NPC, in order to evaluate the value of adjuvant chemotherapy in nasopharyngeal carcinoma (NPC) patients.

DETAILED DESCRIPTION:
Patients presented with non-keratinizing NPC and stage T3-4N1M0/TxN2-3M0 are randomly assigned to receive concurrent chemoradiotherapy plus adjuvant chemotherapy (investigational arm)or concurrent chemoradiotherapy (control arm). Patients in both arms receive radical radiotherapy and cisplatin (40mg/m2 on day 1) weekly during radiotherapy. Patients in the investigational arm receive cisplatin (80mg/m2 on day 1) and fluorouracil (800mg/m2 on Day 1 to 5) every four weeks for three cycles after completion of radiotherapy. Patients are stratified according to the treatment centers. The primary end point was failure-free survival (FFS). Secondary end points included overall survival (OS), distant failure-free survival (D-FFS), locoregional failure-free survival (LR-FFS), the initial response rates after treatments, toxic effects and treatment compliance. All efficacy analyses were conducted in the intention-to-treat population; the safety population included only patients who received their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing carcinoma (according to World Health Organization (WHO) histologically type)
2. Tumor staged as N2-3or T3-4N1 (according to 6th American Joint Committee on Cancer staging system)
3. No evidence of distant metastasis (M0)
4. Performance status: KPS ≥70
5. With normal liver function test (Alanine Aminotransferase、Aspartate Aminotransferase ≤2.5×upper limit of normal)
6. Renal: creatinine clearance ≥60ml/min
7. Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥80g/L and platelet count ≥100000/μL
8. Written informed consent

Exclusion Criteria:

1. WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
2. Age ≥70 or <18
3. With a history of renal disease
4. Prior malignancy
5. Previous chemotherapy or radiotherapy
6. Patient is pregnant or lactating
7. Unstable cardiac disease requiring treatment.
8. Emotion disturbance

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2006-06; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 2-yr
  Failure-free survival is calculated from the date of randomization to the date of the first failure at any site.

SECONDARY OUTCOMES:
Overall survival, distant failure-free survival and locoregional failure-free survival | 2-yr
  Overall survival is calculated from randomization to death from any cause. For distant failure-free survival and locoregional failure-free survival analyses, the latencies to the first remote or local failure, respectively, are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chua DT, Sham JS, Kwong DL, Au GK. Treatment outcome after radiotherapy alone for patients with Stage I-II nasopharyngeal carcinoma. Cancer. 2003 Jul 1;98(1):74-80. doi: 10.1002/cncr.11485. PMID 12833458
- [Background] Ma J, Mai HQ, Hong MH, Cui NJ, Lu TX, Lu LX, Mo HY, Min HQ. Is the 1997 AJCC staging system for nasopharyngeal carcinoma prognostically useful for Chinese patient populations? Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1181-9. doi: 10.1016/s0360-3016(01)01537-1. PMID 11483327
- [Background] Zhao C, Han F, Lu LX, Huang SM, Lin CG, Deng XW, Lu TX, Cui NJ. [Intensity modulated radiotherapy for local-regional advanced nasopharyngeal carcinoma]. Ai Zheng. 2004 Nov;23(11 Suppl):1532-7. Chinese. PMID 15566674
- [Background] Lee N, Xia P, Quivey JM, Sultanem K, Poon I, Akazawa C, Akazawa P, Weinberg V, Fu KK. Intensity-modulated radiotherapy in the treatment of nasopharyngeal carcinoma: an update of the UCSF experience. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):12-22. doi: 10.1016/s0360-3016(02)02724-4. PMID 12007936
- [Background] Kam MK, Teo PM, Chau RM, Cheung KY, Choi PH, Kwan WH, Leung SF, Zee B, Chan AT. Treatment of nasopharyngeal carcinoma with intensity-modulated radiotherapy: the Hong Kong experience. Int J Radiat Oncol Biol Phys. 2004 Dec 1;60(5):1440-50. doi: 10.1016/j.ijrobp.2004.05.022. PMID 15590175
- [Background] Decker DA, Drelichman A, Al-Sarraf M, Crissman J, Reed ML. Chemotherapy for nasopharyngeal carcinoma. A ten-year experience. Cancer. 1983 Aug 15;52(4):602-5. doi: 10.1002/1097-0142(19830815)52:43.0.co;2-6. PMID 6683121
- [Background] Al-Sarraf M. Chemotherapeutic management of head and neck cancer. Cancer Metastasis Rev. 1987;6(3):181-98. doi: 10.1007/BF00144263. PMID 3319271
- [Background] Rossi A, Molinari R, Boracchi P, Del Vecchio M, Marubini E, Nava M, Morandi L, Zucali R, Pilotti S, Grandi C, et al. Adjuvant chemotherapy with vincristine, cyclophosphamide, and doxorubicin after radiotherapy in local-regional nasopharyngeal cancer: results of a 4-year multicenter randomized study. J Clin Oncol. 1988 Sep;6(9):1401-10. doi: 10.1200/JCO.1988.6.9.1401. PMID 3047335
- [Background] Chi KH, Chang YC, Guo WY, Leung MJ, Shiau CY, Chen SY, Wang LW, Lai YL, Hsu MM, Lian SL, Chang CH, Liu TW, Chin YH, Yen SH, Perng CH, Chen KY. A phase III study of adjuvant chemotherapy in advanced nasopharyngeal carcinoma patients. Int J Radiat Oncol Biol Phys. 2002 Apr 1;52(5):1238-44. doi: 10.1016/s0360-3016(01)02781-x. PMID 11955734
- [Background] Frederick L. Greene, David L. Page, Irvin D. Fleming, et al: American Joint Committee on Cancer Staging Manual (ed 6). Philadelphia (PA): Lippincott, 2002.
- [Background] Freedman J, Furberg, C, DeMets D. Fundamentals of clinical trials. Springer-Verlag, NY, 1998.
- [Background] Chow, S.C., Shao, J., Wang, H. Sample Size Calculations in Clinical Research. New York: Marcel Dekker; 2003.
- [Derived] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Adjuvant chemotherapy in patients with locoregionally advanced nasopharyngeal carcinoma: Long-term results of a phase 3 multicentre randomised controlled trial. Eur J Cancer. 2017 Apr;75:150-158. doi: 10.1016/j.ejca.2017.01.002. Epub 2017 Feb 22. PMID 28235726
- [Derived] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591